CLINICAL TRIAL: NCT07160231
Title: REDO-JAK: Dose REDuction Of JAnus Kinase Inhibitors in Patients With Inflammatory Rheumatic Diseases
Acronym: REDO-JAK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1172; 2025-520757-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA); Psoriatic Arthritis (PsA); Axial Spondyloarthritis (AxSpA)
Keywords: disease activity guided dose reduction; Janus kinase inhibitors (JAKi); disease activity guided JAKi continuation
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: This open label study is a partially randomised patient preference trial (PRPPT), also known as comprehensive cohort study (CCS). The PRPPT design includes two subtrials that will subsequently be pooled to derive a single treatment effect estimate. The first is a pragmatic randomised controlled trial including participants who consent to randomisation. In addition, a non-randomised trial is done using the same intervention, control arm and outcome assessments, but allocation based on patient preferences.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Dose reduction group (randomised) (Experimental): disease activity guided dose reduction strategy of JAKi
  Interventions: Drug: JAKi dose reduction strategy
- Control group (randomised) (Active Comparator): disease activity guided continuation of same dose strategy of JAKi (randomised)
  Interventions: Drug: JAKi disease activity guided continuation of same dose strategy
- Dose reduction group (non-randomised) (Experimental): disease activity guided dose reduction strategy of JAKi
  Interventions: Drug: JAKi dose reduction strategy
- Control group (non-randomised) (Active Comparator): disease activity guided continuation of same dose strategy of JAKi
  Interventions: Drug: JAKi disease activity guided continuation of same dose strategy

INTERVENTIONS:
Drug: JAKi dose reduction strategy — JAKi dose reduction strategy
  Arms: Dose reduction group (non-randomised); Dose reduction group (randomised)
Drug: JAKi disease activity guided continuation of same dose strategy — JAKi disease activity guided continuation of same dose strategy
  Arms: Control group (non-randomised); Control group (randomised)

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of a disease activity guided dose reduction strategy of Janus kinase inhibitor (JAKi) compared to disease activity guided JAKi continuation in patients with rheumatoid arthritis (RA), psoriatic arthritis (PsA) and axial spondyloarthritis (axSpA) who are in a state of low disease activity or remission while on JAKi. The main question it aims to answer is:

Is a disease activity guided dose reduction strategy for JAKi not inferior in terms of efficacy compared to disease activity guided JAKi continuation in patients with RA/PsA/axSpA that are currently in a low disease activity/remission state?

Researchers will compare a disease activity guided dose reduction strategy for JAKi to disease activity guided JAKi continuation in patients with RA/PsA/axSpA that are currently in a low disease activity/remission state to see if a disease activity guided dose reduction strategy for JAKi is not inferior in terms of efficacy compared to disease activity guided JAKi continuation.

Participants will:

* Follow a JAKi dose reduction strategy or will continue using JAKi in the same dose
* Study (telemonitoring) visits are planned every 3 months
* At every visit, patients are asked to complete patient-reported outcomes that assess daily functioning, health-related quality of life, pain, fatigue, productivity loss, medical consumption and medication adherence.

DETAILED DESCRIPTION:
Rationale Janus kinase inhibitors (JAKi) are used in the treatment of rheumatoid arthritis (RA), psoriatic arthritis (PsA), and axial spondyloarthritis (axSpA). Despite their proven effectiveness, use of these drugs increases the risk of infections and is costly. In addition, there have been recent warnings that JAKi may increase the risk of cardiovascular disease and cancer. For other anti-rheumatic drugs, disease activity guided dose reduction has been shown to be safe and cost-effective while reducing side effects. This has not yet been studied for JAK inhibitors, while it is very relevant given the concerns regarding side effects and costs of the drugs.

Objective The primary objective of this project is to assess the effectiveness of a disease activity guided dose reduction strategy of JAKi compared to disease activity guided JAKi continuation in patients with RA, PsA and axSpA who are in a state of low disease activity or remission while on JAKi. Key secondary objectives are to assess feasibility of the proposed dose reduction strategies, safety, cost-effectiveness and the identification of possible predictive biomarkers for (un)successful dose reduction or discontinuation of JAKi.

Main trial endpoints The main trial endpoint is the non-inferiority of the difference in the proportion of people with low disease activity between the dose reduction group and the continuation group after 12 months compared to the non-inferiority margin.

Secondary trial endpoints Secondary trial endpoints include the proportion of people in the intervention group able to reduce and/or discontinue their JAKi, cost-effectiveness of the dose reduction strategy compared to the continuation strategy, and between group differences in the incidence of disease flares, difference in functioning, quality of life, pain, fatigue, safety and costs.

Trial design This open label study is a partially randomised patient preference trial, also known as a comprehensive cohort study. Participants will be randomised (2:1 ratio) to step-by-step dose reduction or continuation of standard dosing. If potential participants have a strong preference for a specific group and do not wish to be randomised, they will be given the opportunity to choose their group. Follow up for and individual patient is this trial will be 12 months.

Trial population Patients ≥ 16 year, with a clinical diagnosis of RA, PsA or axSpA who use a JAK inhibitor and have low disease activity.

Interventions The intervention group reduces their JAKi dose stepwise every three months. In the event of a flare of disease activity, the dose is increased to the latest effective dose and kept stable until the end of follow-up.

A dose reduction scheme is created for each JAKi for patients allocated to the intervention group:

For patients using:

Baricitinib 4 mg once daily Dose reduction step 1 (baseline); 2 mg once daily (splitting 4 mg tablet) Dose reduction step 2 (3 months); 1 mg once daily (splitting 2 mg tablet) Dose reduction step 3 (6 months); Discontinuation

Baricitinib 2 mg once daily Dose reduction step 1 (baseline) 1 mg once daily (splitting 2 mg tablet) Dose reduction step 2 (3 months); Discontinuation

Filgotinib 200 mg once daily Dose reduction step 1 (baseline); 100 mg once daily (splitting 200 mg tablet) Dose reduction step 2 (3 months); 50 mg once daily (splitting 100 mg tablet) Dose reduction step 3 (6 months); Discontinuation

Filgotinib 100 mg once daily Dose reduction step 1 (baseline); 50 mg once daily (splitting 100 mg tablet) Dose reduction step 2 (3 months); Discontinuation

Tofacitinib 5 mg twice daily OR Tofacitinib 11 mg once daily Dose reduction step 1 (baseline); 5 mg once daily Dose reduction step 2 (3 months); 2.5 mg once daily (splitting 5mg tablet) Dose reduction step 3 (6 months); Discontinuation

Tofacitinib 5 mg once daily Dose reduction step 1 (baseline); 2.5 mg once daily (splitting 5mg tablet) Dose reduction step 2 (3 months); Discontinuation

Upadacitinib 15 mg once daily Dose reduction step 1 (baseline); 7.5 mg once daily (splitting 15 mg tablet) Dose reduction step 2 (3 months); 7.5 mg every other day (splitting 15 mg tablet) Dose reduction step 3 (6 months); Discontinuation

The control group continues treatment following usual care. All participants are monitored every 3 months. For both trial arms, additional visits can be scheduled in between planned visits in case of complaints. In case of flare treatment will be intensified.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 16 years of age
* Clinical diagnosis of RA, PsA or axSpA
* Treated with a JAKi (monotherapy or combination with csDMARDwith a JAKi dose ≥ 50% of the authorised dose)
* LDA or remission for at least 6 months according to accepted criteria for the specific disease and/or the judgement of the treating rheumatologist and patient. (RA: DAS28-CRP < 2.9; PsA: PASDAS ≤3.2 and psoriasis mBSA involvement ≤3%; axSpA: ASDAS <2.1.)

Exclusion Criteria:

* Comorbidity for which continued JAKi treatment is expected to be necessary (e.g. active Crohn's disease, ulcerative colitis)
* Life expectancy ≤12 months
* Pregnancy (JAKi are contra-indicated during pregnancy, therefore we do not expect patients using a JAKi while pregnant)
* Patients who are enrolled in other trials that might mutually interfere
* Not able to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients in low disease activity (LDA) at 12 months of follow-up in each study group. | At 12 months of follow-up.
  The proportion of patients in low disease activity (LDA) at 12 months of follow-up in each study group. LDA is defined as DAS28-CRP < 2.9 for RA patients, PASDAS < 3.2 and mBSA involvement ≤3% for PsA and ASDAS < 2.1 and an absence of active extra musculoskeletal symptoms for axSpA.

SECONDARY OUTCOMES:
Mean DAS28-CRP for RA patients, PASDAS for PsA patients and ASDAS for AxSpA patients. | At 6 and 12 months of follow up.
  Mean DAS28-CRP for RA patients, PASDAS for PsA patients and ASDAS for AxSpA patients at 6 and 12 months of follow up in each study group.
Proportion of patients in intervention group at every dose reduction step. | At 6 and 12 months of follow up.
  Proportion of patients in intervention group at every dose reduction step (including discontinuation) at 6 and 12 months of follow up.
The proportion of patients developing adverse events in each study group. | Through study completion, an average of 12 months
  The proportion (cumulative incidence and incidence density) of patients developing (treatment-related) adverse events in each study group over the duration of the study, with special attention to infections, anaemia, cardiovascular events, VTE and malignancies.
The cumulative incidence of patients experiencing a flare. | Through study completion, an average of 12 months
  The cumulative incidence of patients experiencing a flare in each study group over the duration of the study.
Proportion of patients using comedication. | At baseline and through study completion, an average of 12 months
  Proportion of patients using csDMARD, corticosteroids or NSAIDs at baseline, and starting/changing these treatments during follow-up.
The incremental cost effectiveness ratio | Through study completion, an average of 12 months
  Quality of life and costs incurred during the study will be compared between the study groups. The incremental cost effectiveness ratio will be calculated using incremental (between-group) costs and quality of life, and compared with different willingness to pay thresholds.
Association between possible predictors and outcome. | Through study completion, an average of 12 months
  Association between possible predictors and outcome. Predictors will include baseline peak and trough JAKi concentrations and whole blood/PBMC immunophenotyping.

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - Sint Maartenskliniek Nijmegen, Nijmegen, Gelderland
  - Maastricht UMC+, Maastricht, Limburg
  - Elisabeth-TweeSteden Ziekenhuis Tilburg, Tilburg, North Brabant
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Isala Zwolle, Zwolle, Overijssel
  - Erasmus MC, Rotterdam, South Holland
  - Maasstad ziekenhuis, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No